CLINICAL TRIAL: NCT03308552
Title: A Randomized Phase III Study of Simultaneous Integrated Boost Intensity Modulated Radiation Therapy (SIB-IMRT) With or Without Concurrent Chemotherapy Followed by Consolidation Chemotherapy for Limited Lymphatic Metastasis of Esophageal Cancer - 3JECROG-P02
Brief Title: Radiotherapy With or Without Concurrent Chemotherapy for Limited Lymphatic Metastasis of Esophageal Cancer - 3JECROG P-02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Anyang Tumor Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Affiliated Hospital of Hebei University (Other); Fujian Cancer Hospital (Other Government); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3JECROG P-02
Record Dates: First submitted 2017-10-08; First posted 2017-10-12 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIB-IMRT combined chemotherapy followed by chemotherapy (Active Comparator): SIB-IMRT: Patients receive radiotherapy once daily, 5 days a week for an average of 5.5 weeks. Radiotherapy is delivered to achieve a prophylactic dosage of 50.4Gy to PTV and 59.92Gy to PGTV in 28 fractions, respectively.
  Concurrent chemotherapy: Paclitaxel and platinum based drug are administered once a week for at least 5 weeks during radiotherapy treatment days.
  Interventions: Radiation: SIB-IMRT; Drug: Paclitaxel; Drug: Platinum-Based Drug
- SIB-IMRT Alone followed by chemotherapy (Placebo Comparator): SIB-IMRT: Patients receive radiotherapy once daily, 5 days a week for an average of 5.5 weeks. Radiotherapy is delivered to achieve a prophylactic dosage of 50.4Gy to PTV and 59.92Gy to PGTV in 28 fractions, respectively.
  Interventions: Radiation: SIB-IMRT; Drug: Paclitaxel; Drug: Platinum-Based Drug

INTERVENTIONS:
Radiation: SIB-IMRT — PTV:50.4Gy/28f, PGTV:59.92Gy/28f
Drug: Paclitaxel — 45-50 mg/m2, once a week, concurrent with radiotherapy for 5-6weeks
  Arms: SIB-IMRT combined chemotherapy followed by chemotherapy
Drug: Platinum-Based Drug — Nedaplatin or Lobaplatin or Cisplatin, 20-25mg/m2, once a week, concurrent with radiotherapy for 5-6weeks
  Arms: SIB-IMRT combined chemotherapy followed by chemotherapy
Drug: Paclitaxel — 150mg/m2 on day1,every 3 weeks, 4 cycles, 1-3 months after completion of radiotherapy
Drug: Platinum-Based Drug — Nedaplatin or Lobaplatin or Cisplatin, 50-80mg/m2 on day1 (Lobaplatin 50mg on day 1),every 3 weeks, 4 cycles, 1 month after completion of radiotherapy

SUMMARY:
This phase III trial is designed to explore a higher radiation dose by using IMRT simultaneous integrated boost technique with or without concurrent chemotherapy for esophageal carcinoma with limited lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Age<70
* Diagnosis of clinical stage T2-4N0-1M1（According to UICC 2002）
* A untreated squamous esophageal carcinoma
* Karnofsky performance status(KPS)≥ 70 and Charlson score ≤3
* Adequate organ function
* No known history of drug allergy
* Blood routine examination : WBC≥4.0
* hepatic and renal function are normal

Exclusion Criteria:

* Age≥ 70 or < 18
* Already received the treatment of chemotherapy or radiotherapy
* Pregnant or lactating females
* Known drug allergy
* Without agreement of informed consent form
* Insufficient hepatorenal function or Blood routine examination
* Severe cardiovascular diseases, diabetes with uncontrolled blood sugar, mental disorders, uncontrolled severe infection, active ulceration which need intervention.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival（OS） | 1 year
Overall survival（OS） | 2 year
Overall survival（OS） | 3 year

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Progress free survival（PFS） | 2 year
Progress free survival（PFS） | 3 year
Local recurrence-free rate（LRFS） | 1 year
Local recurrence-free rate（LRFS） | 2 year
Local recurrence-free rate（LRFS） | 3 year
Completion Rate | up to 2 year
  the completion rate of each arm
Adverse events | up to 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, MD, Principal Investigator — The Department of Radiation Oncology ,Cancer Institute & Hospital，Chinese Academy of Medical Science
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao LR, Wang X, Han W, Deng W, Li C, Wang X, Zhao Y, Ni W, Chang X, Zhou Z, Deng L, Wang W, Liu W, Liang J, Zhang T, Bi N, Wang J, Zhai Y, Feng Q, Lv J, Li L, Xiao Z. A multicenter prospective phase III clinical randomized study of simultaneous integrated boost intensity-modulated radiotherapy with or without concurrent chemotherapy in patients with esophageal cancer: 3JECROG P-02 study protocol. BMC Cancer. 2020 Sep 22;20(1):901. doi: 10.1186/s12885-020-07387-y. PMID 32962674